CLINICAL TRIAL: NCT00710619
Title: Dosing Observational Study in Hemophilia Subjects With Inhibitors: A Phase IV Diary Study in Subjects Prescribed NovoSeven® as First Line on Demand Therapy for Acute Bleeding Episodes
Brief Title: Observational Patient Diary Study of Treatment Doses for Patients With Haemophilia With Inhibitors to Factors VIII and IX
Acronym: DOSE
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: F7HAEM-1965
Record Dates: First submitted 2008-07-03; First posted 2008-07-04 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2016-11

CONDITIONS: Congenital Bleeding Disorder; Haemophilia A With Inhibitors; Haemophilia B With Inhibitors
MeSH Terms: interventions — anti-inhibitor coagulant complex

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Drug: activated recombinant human factor VII; Drug: Feiba VH

INTERVENTIONS:
Drug: activated recombinant human factor VII — This is an observation of how patients/caregivers dose bypassing agents at home for haemophilia with inhibitors
Drug: Feiba VH — This is an observation of how patients/caregivers dose bypassing agents at home for hemophilia with inhibitors

SUMMARY:
This study is conducted in the United States of America (USA). The aim of this study is to investigate the at-home-administration of bypassing agents for treatment of bleeding episodes in patients with congenital haemophilia with inhibitors to factors VIII and IX. We are further investigating how bleeding episodes affect the quality of life of the patient and their family or caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects with congenital haemophilia A or B and inhibitors with spontaneous bleeds which require on-demand treatment
* Subjects prescribed NovoSeven® as the first line or recommended bypass agent
* History of on average at least 4 bleeds of any type over a 3 month period
* Subject or caregiver able and willing to complete daily journal for 3 months
* Informed consent obtained from all subjects or legal representative

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male subjects with congenital haemophilia A or B with inhibitors with spontaneous bleeds requiring on-demand treatment
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2008-06; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Characterisation of dose and dosing intervals for each bleeding episode | after 3-6 months

SECONDARY OUTCOMES:
Effect of type of bleed on initial dose, dosing interval and total dose | after 3-6 months
Effect of initial dose and dosing interval on total dose, time to first perceived improvement, time to perceived bleed resolution | after 3-6 months
Effect of time to first dose on dosing interval and total dose | after 3-6 months
Effect of bleeds and drug administration time on planned daily activities | after 3-6 months
Relationship of dose and dosing intervals to reported SAEs | after 3-6 months

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Plainsboro, New Jersey, United States

REFERENCES:
- [Derived] Gruppo RA, Kessler CM, Neufeld EJ, Cooper DL. Assessment of individual dose utilization vs. physician prescribing recommendations for recombinant activated factor VII (rFVIIa) in paediatric and adult patients with congenital haemophilia and alloantibody inhibitors (CHwI): the Dosing Observational Study in Hemophilia (DOSE). Haemophilia. 2013 Jul;19(4):524-32. doi: 10.1111/hae.12113. Epub 2013 Apr 1. PMID 23551918
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com